CLINICAL TRIAL: NCT01107574
Title: Phase III Study of the Use of Gabapentin and Osteopathic Manipulative Medicine to Treat Fibromyalgia
Brief Title: Fibromyalgia Treatment Trial With Gabapentin and Osteopathic Manipulative Medicine
Acronym: FTTGO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Good Samaritan Regional Medical Center, Oregon (Other)
Collaborators: Touro University,Vallejo,California (Unknown)
Responsible Party: Principal Investigator, Cynthia S. Marske DO, Program Director Internal Medicine Residency, Good Samaritan Regional Medical Center, Oregon
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-01-2004
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Fibromyalgia
Keywords: Chronic Pain, tenderpoints, insomnia, mood disorder, fatigue
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Sleep Initiation and Maintenance Disorders; Mood Disorders; Fatigue | interventions — Gabapentin; Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gabapentin and Osteopathic Manipulative Medicine (Experimental): 6 weeks of both Gabapentin 900 mg HS given orally was accompanied with Osteopathic Manipulative Medicine treatment 30 minutes weekly to the tender points of the musculoskeletal system of each patient for 6 weeks.
  Interventions: Other: Gabapentin and Osteopathic Manipulative Medicine
- Gabapentin (Experimental): Gabapentin was given orally at 900 mg at HS weekly for 6 weeks.
  Interventions: Drug: Gabapentin
- Osteopathic Manipulative Medicine (Experimental): 6 weeks of Osteopathic Manipulative Medicine Treatment was applied to the patients tender points in the musculoskeletal system weekly by a 30 minute treatment.
  Interventions: Procedure: Osteopathic Manipulative Medicine

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 900 mg po HS for 6 weeks treatment per patients enrolled in the Gabapentin Arm
  Other Names: Neurontin
  Arms: Gabapentin
Procedure: Osteopathic Manipulative Medicine — Based on Osteopathic Structural Examination and Tender point Examination a 30 minute treatment of Osteopathic Manipulative Medicine was applied to each patient every week for 6 weeks.
  Other Names: Osteopathic Manipulation Treatment
  Arms: Osteopathic Manipulative Medicine
Other: Gabapentin and Osteopathic Manipulative Medicine — Combination therapy of gabapentin 900 mg po HS for 6 weeks and Osteopathic Manipulative Medicine 30 minute treatment weekly for each patient based on Osteopathic Structural Examination and Tender point Examination
  Other Names: Combined OMM and Neurontin
  Arms: Gabapentin and Osteopathic Manipulative Medicine

SUMMARY:
This study assesses the benefits of intervention with gabapentin, Osteopathic Manipulative Medicine or both for improvement of the symptoms of Fibromyalgia. This study also seeks to determine whether these treatments will decrease the number and severity of tender points, improve structure, function and the overall pain level of each patient from the baseline of the study to the end. This study is designed to evaluate whether subjects subjectively experience an improved quality of life and increased function as a result of these interventions corresponding to objective improvements.

DETAILED DESCRIPTION:
An 8-week, randomized, study was designed to compare gabapentin (900 mg/day) (n = 8 patients) with OMM (n = 11 patients) with Combined treatment of gabapentin (900 mg/day) plus OMM (n = 7 patients) for efficacy and safety in treating pain, fatigue, depression and function associated with fibromyalgia.

The primary outcome measures were measured during week 2 and week 8 to evaluate efficacy of each arm and compare efficacy between each arm at improving structure, function and pain. The Baker Wong Brief Pain Inventory (BPI) was evaluated weekly for average pain severity score (range 0-10, where 0 = no pain and 10 = pain as bad as you can imagine). Fibromyalgia Impact Questionnaire (FIQ) a tool that evaluates function and health status was administered at week 2 and week 8 for comparison of functioning at the baseline and end of the study. The total number of Tender Points (0-18) as determined by the American College of Rheumatology was counted at week 2 and week 8 to compare number of tender points from the baseline to the end. Dolorimetry in Kg/cm2 as measured by the Fischer Dolorimeter were measured on the 4 most severe tender points at week 2 and week 8 to compare severity of tender points from baseline to end of study. The Osteopathic Structural Examination which measures free range of motion of joints in degrees was measured with goniometry at week 2 and week 8 to evaluate degrees of free range of motion improved from baseline. The Clinical Global Impression which is a likert scale of 1-5 asking patients to evaluate how they feel about their overall health was taken at week 2 and week 8 to see if overall subjective thoughts of health were improved from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients were eligible for the study if they were 18-65 years of age and met the ACR criteria for fibromyalgia ([1]).

Exclusion Criteria:

* Patients with other rheumatic or medical disorders that contributed to the symptoms of fibromyalgia were excluded.
* Rheumatoid arthritis, inflammatory arthritis, or autoimmune disease;
* Pain from traumatic injury or structural or regional rheumatic disease;
* Rheumatoid arthritis, inflammatory arthritis, or autoimmune disease;
* Unstable medical or psychiatric illness;
* Lifetime history of psychosis, hypomania or mania, epilepsy, or dementia;
* Substance abuse in the last 6 months;
* Serious risk of suicide;
* Pregnancy or breastfeeding;
* Unacceptable contraception in those of childbearing potential;
* Patients who, in the opinion of the investigator, were treatment refractory; and prior failed treatment with gabapentin, pregabalin or OMM.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-04; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Outcomes of Efficacy and Tolerability by measure of scored visual tools | 8 Weeks
  Efficacy by Wong-Baker Pain Scale, Fibromyalgia Impact questionaire,Osteopathic Structural Exam, Clinical Global Impression of Change, Tenderpoints and Dolorimetry were assessed at week one and week 8 of treatment.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 8 weeks
  safety of Osteopathic Manipulative Medicine and Gapapentin by evaluation of treatment reactions weekly and laboratories before and after the study.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gugliucci, MD, PhD, Study Director — Touro University-CA, Vallejo
Locations (1):
- Touro University College of Osteoapathic Medicine, Vallejo, California, United States

REFERENCES:
- [Background] Antai-Otong D. The art of prescribing. Depression and fibromyalgia syndrome (FMS): pharmacologic considerations. Perspect Psychiatr Care. 2005 Jul-Sep;41(3):146-8. doi: 10.1111/j.1744-6163.2005.00028.x. No abstract available. PMID 16138826
- [Background] Arnold LM, Goldenberg DL, Stanford SB, Lalonde JK, Sandhu HS, Keck PE Jr, Welge JA, Bishop F, Stanford KE, Hess EV, Hudson JI. Gabapentin in the treatment of fibromyalgia: a randomized, double-blind, placebo-controlled, multicenter trial. Arthritis Rheum. 2007 Apr;56(4):1336-44. doi: 10.1002/art.22457. PMID 17393438
- [Background] Bennett RM. Emerging concepts in the neurobiology of chronic pain: evidence of abnormal sensory processing in fibromyalgia. Mayo Clin Proc. 1999 Apr;74(4):385-98. doi: 10.4065/74.4.385. PMID 10221469
- [Background] Blunt KL, Rajwani MH, Guerriero RC. The effectiveness of chiropractic management of fibromyalgia patients: a pilot study. J Manipulative Physiol Ther. 1997 Jul-Aug;20(6):389-99. PMID 9272472
- [Background] Gamber RG, Shores JH, Russo DP, Jimenez C, Rubin BR. Osteopathic manipulative treatment in conjunction with medication relieves pain associated with fibromyalgia syndrome: results of a randomized clinical pilot project. J Am Osteopath Assoc. 2002 Jun;102(6):321-5. PMID 12090649
- [Background] Hains G, Hains F. A combined ischemic compression and spinal manipulation in the treatment of fibromyalgia: a preliminary estimate of dose and efficacy. J Manipulative Physiol Ther. 2000 May;23(4):225-30. PMID 10820294
- [Background] Johnson SM, Kurtz ME. Osteopathic manipulative treatment techniques preferred by contemporary osteopathic physicians. J Am Osteopath Assoc. 2003 May;103(5):219-24. PMID 12776762
- [Background] Maizels M, McCarberg B. Antidepressants and antiepileptic drugs for chronic non-cancer pain. Am Fam Physician. 2005 Feb 1;71(3):483-90. PMID 15712623
- [Background] McCleane G. Gabapentin reduces chronic benign nociceptive pain: a double-blind, placebo-controlled cross-over study. The Pain Clinic. 2000; 12(2):81-85.
- [Background] Noller V, Sprott H. Prospective epidemiological observations on the course of the disease in fibromyalgia patients. J Negat Results Biomed. 2003 Aug 23;2:4. doi: 10.1186/1477-5751-2-4. PMID 12969513
- [Background] Rivera J, Gonzalez T. The Fibromyalgia Impact Questionnaire: a validated Spanish version to assess the health status in women with fibromyalgia. Clin Exp Rheumatol. 2004 Sep-Oct;22(5):554-60. PMID 15485007
- [Background] Hansen HC. Treatment of chronic pain with antiepileptic drugs: a new era. South Med J. 1999 Jul;92(7):642-9. doi: 10.1097/00007611-199907000-00001. PMID 10414471
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- See also: Department of Research — http://www.tu.edu